## <u>Community Development and Nutrition Education in Banke District, Nepal: Effect on Child Health and Growth</u>

Today's date: April 20, 2018

Date of Approval of Study Protocol by Tufts IRB: October 2, 2014

NCT: not yet available

## **Study protocol**

Throughout Nepal, small community organizations approach Heifer to request inputs. Because of high demand for these inputs, Heifer responds to these requests sequentially. For this investigation, similar community organizations (all located in the Banke district of Nepal) which have requested Heifer inputs will be matched based on specific characteristics, including size, altitude, income profiles, type of agriculture practiced, current livestock inventories, availability of medical services, family size, household income, castes, feeding practices, local natural resources (e.g., fresh water, wood for fuel, etc.), educational level of adult community members, nutritional status of children, and known local health risks (e.g. lead exposure, iodine deficiency). Leaders of these community organizations will be informed about the project and invited to participate. Matched clusters of households willing to participate will be identified and randomly assigned to one of three arms of the investigation: (1) Full Heifer inputs (including training in social capital, community development, livestock management, and nutrition), (2) livestock management and nutrition training only, or (3) control group. After the investigation is complete, the Control group communities will receive full Heifer inputs (training in social capital, community development, livestock management, and nutrition) and the Training Only Group will receive social capital and community development training. Thus, all communities will receive the complete package of Heifer social capital, community development, livestock management, and nutrition training; only the timing for these activities will be altered to allow the study of suitable comparison groups.

Data collection methods. Trained field enumerators will visit each household every 6 months for 2 years (total 5 visits: baseline, 6 months, 12 months, 18 months and 24 months). At each visit, a questionnaire will be administered to the mother in the household or the household head (estimated 1 hr completion). All children from ages 1 month to 7 yrs 11 months will be weighed, and height, head circumference, and mid upper-arm circumference will be measured. Thus, mothers (or household head) and children in the target age range will be research participants.